CLINICAL TRIAL: NCT01348789
Title: Safety of Hair2Go Device in Frequent Use Conditions: A Prospective, Open Label Study With Before-After Design
Brief Title: Safety for Frequent Use Conditions of Hair Removal Device
Acronym: OHR-3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Syneron Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OHR-3
Record Dates: First submitted 2011-05-04; First posted 2011-05-05 (Estimated); Results first posted 2013-02-18 (Estimated); Last update posted 2013-02-18 (Estimated); Status verified 2013-02

CONDITIONS: Hair Removal
Keywords: Hair removal; Hair Clearance; Epilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Hair2Go (Mē) (Experimental): Treatment with Hair2Go (Mē)device
  Interventions: Device: Hair2Go (Mē)

INTERVENTIONS:
Device: Hair2Go (Mē) — Treatment with Hair2Go (Mē) three times every 2-4 days
  Other Names: Mē my elōs

SUMMARY:
To measure the safety of hair removal device when used frequently.

DETAILED DESCRIPTION:
The primary endpoint of this study is to measure the safety of the Hair2Go device when used frequently. The secondary endpoints include the kinetics of the hair clearance up to 8 weeks after the last treatment, and gathering information about the pain associated with the procedure

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females, between 18 and 65 years of age.
* Willing to sign informed consent.
* Willing to follow the treatment schedule and post treatment follow-up.
* Willingness to have photographs of the treated area taken that may be used for marketing and educational presentation and/or publications
* Willingness to avoid excessive sun exposure two weeks prior treatments

Exclusion Criteria:

* A history of keloidal scarring (hypertrophic scars or keloids).
* Active dermatologic lesion or infection in the treatment site.
* Subject has permanent tattoos or makeup in the treatment area.
* Recently tanned in the area to be treated and/or unable or unlikely to refrain from tanning during the study.
* Subject has disease related to photosensitivity, such as porphyria, polymorphic light eruption, solar urticaria, lupus, etc
* Subject has a history of herpes outbreak in the area of treatment, unless receiving preventative treatment from physician
* Pregnant, planning to become pregnant, hormone fluctuations and/or breast feeding during the experiment.
* Subjects with Diabetes (Type I or II) or other systemic or metabolic condition
* Subject has an active electrical implant anywhere in the body, such as a pacemaker, an internal defibrillator, insulin pump, incontinence device, etc.
* Subject suffers from epilepsy.
* Subject has active cancer, or has a history of skin cancer or any other cancer in the area to be treated, including presence of malignant or pre-malignant pigmented lesions.
* Subject received radiation therapy or chemotherapy treatments with the past 3 months.
* Subject has known anticoagulative or thromboembolic condition or is on any form of anticoagulation treatment.
* Subject has a history of immunosuppressant/immune deficiency disorders (including HIV infection or AIDS) or currently using immunosuppressive medications.
* Subject has any other condition which in the physician's opinion would make it unsafe for the subject to be treated.
* Subject had rotating type tweezer epilator treatment, or waxing within the last 3 months
* Subject had electrolysis treatment within the last 6 months over the treatment area.
* Subject had any type of professional intense pulsed light (IPL), laser or RF hair removal in the treatment site within the last 6 months.
* Participation in a study of another device or drug within 1 month prior to enrollment or during this study.
* Subject is taking medication known to induce photosensitivity, including non-steroidal anti-inflammatory agents, tetracyclines, phenothiazines, thiazide diuretics, sulfonylureas, sulfonamides, Dacarbazine (DTIC), fluorouracil, vinblastine, and griseofulvin within 4 weeks of therapy.
* Subject has been taking Accutane® within 6 months of therapy.
* Subject has been on steroid regimen during the last three months.
* Subject is on Gold therapy (for arthritis treatment).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2011-03; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jerome M Garden, MD, Principal Investigator — Northwestern Memorial Hospital
Locations (1):
- Physician Laser and Dermatology Institute, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment was conducted in a medical clinic. The recruitment continued from January to June 2011.
Groups:
- Hair2Go (Mē): Treatment with Hair2Go (Mē)device - 3 treatments in 2-4 day intervals
Period: Overall Study
Arm/Group | Hair2Go (Mē)
Started | 37
Completed | 33 (4 subjects did not complete all 3 treatments but were evaluated for primary and secondary endpoints.)
Not Completed | 4
Not completed — Protocol Violation | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Hair2Go (Mē)
Number analyzed (Participants) | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 37
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 32.5 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 37

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Device Related Anticipated Skin Effects, Serious Adverse Events, or Adverse Events.
Description: The immediate skin reaction and long-term side and adverse effects were evaluated on site by a dermatologist. This includes the following clinical outcomes:
  * Presence of transient (disappearing < 24 hours) or prolonged erythema
  * Presence of transient (disappearing < 24 hours) or prolonged edema
  * Self-limited bleeding from mechanical shaving
  * Blister formation
  * Ulcer formation
  * Pigment changes (hypo/hyper)
  * Textural changes
  * Scarring
  * Infection
  * Pruritis
  * Post inflammation reactions
  * Allergic reaction
  The safety of the device will be confirmed if no device related serious adverse event will occur.
Time Frame: Up to 3 months
Population: Intention to treat analysis - all participants that received at least 1 treatment.
Measure: Number (95% Confidence Interval); unit: percentage of particpants
Arm/Group | Hair2Go (Mē)
Number analyzed (Participants) | 37
percentage of particpants
  Anticipated skin effects | 0 [0 to 9.5]
  Device related serious adverse events | 0 [0 to 0.83]
  Device related adverse events | 0 [0 to 9.5]

2. Secondary Outcome: Tolerability Level of the Procedure for Each Treatment Separately for Light and Dark Skin.
Description: Subject self-report of the tolerability of the procedure (no pain, mild pain, moderate pain) after each of the treatments (#1, #2, #3)separately for relatively light and dark skin photo-types (I-IV and V-VI respectively according to Fitzpatrick skin photo-type classification)
Time Frame: 0, 3, 7 days (after treatment #1, #2, and #3 respectively)
Measure: Number; unit: number of areas
Units Other Than Participants: Treatment areas
Groups:
- Light Skin - Treat#1: Self assessment of tolerability for skin photo-type I-IV after treatment#1.
- Light Skin - Treat#2: Self assessment of tolerability for skin photo-type I-IV after treatment#2.
- Light Skin - Treat#3: Self assessment of tolerability for skin photo-type I-IV after treatment#3.
- Dark Skin - Treat#1: Self assessment of tolerability for skin photo-type V-VI after treatment#1
- Dark Skin - Treat#2: Self assessment of tolerability for skin photo-type V-VI after treatment#2
- Dark Skin - Treat#3: Self assessment of tolerability for skin photo-type V-VI after treatment#3
Arm/Group | Light Skin - Treat#1 | Light Skin - Treat#2 | Light Skin - Treat#3 | Dark Skin - Treat#1 | Dark Skin - Treat#2 | Dark Skin - Treat#3
Number analyzed (Participants) | 20 | 19 | 16 | 17 | 17 | 17
Number analyzed (Treatment areas) | 86 | 82 | 70 | 68 | 68 | 68
number of areas
  No Pain | 82 | 80 | 70 | 50 | 53 | 54
  Mild pain | 4 | 2 | 0 | 13 | 13 | 12
  Moderate Pain | 0 | 0 | 0 | 5 | 2 | 2

3. Secondary Outcome: Hair Clearance
Description: Hair Clearance = the percent of hair cleared from baseline to follow up
Time Frame: 8 weeks after last treatment
Measure: Median (Standard Deviation); unit: %baseline hair count
Units Other Than Participants: Treated areas
Groups:
- Hair Clearance From All Areas: Treatment with Hair2Go (Mē) device
Arm/Group | Hair Clearance From All Areas
Number analyzed (Participants) | 37
Number analyzed (Treated areas) | 71
%baseline hair count | 44.19 (31.09) [37.1 to 51.3]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Hair2Go (Mē)
Serious Adverse Events (participants affected / at risk) | 0/37
Other Adverse Events (participants affected / at risk) | 0/37

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days